CLINICAL TRIAL: NCT06912464
Title: Comparative Safety Analysis: PET vs. CT Scans During Intensive Care Admission
Brief Title: To Evaluate Transport Safety Between Different Scanning Methods for Patients in the Intensive Care Unit (ICU)
Acronym: CASA
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 20649
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Transportation of Patients; PET / CT; Intensive Care Medicine
Keywords: Intrahospital transport (IHT); Intensive Care Medicine; ICU; PET; PET/CT; Safety; CT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PET/CT: Patients undergoing a PET/CT for any reason will be evaluated for safety.
- CT: All patients undergoing a (planned) CT-Thorax/Abdomen will be included in the analysis.

SUMMARY:
The goal of this study is to assess how safe it is for critically ill patients in the Intensive Care Unit (ICU) to undergo a PET scan. A PET scan is a type of medical imaging used to help determine why a patient is sick. It is similar to a CT scan but involves a small amount of radioactivity to highlight areas of concern in the body.

For a PET scan, patients need to be transported from the ICU to the scanning room, which can be risky because ICU patients are often very fragile. After a patient gets the PET scan injection, their body gives off a small amount of radiation for a short time. Because of this, doctors and nurses have to keep some distance to protect themselves. This means they keep an eye out for the patient from a bit further away than normal. This makes the procedure slightly riskier, especially for very sick patients.

This study aims to answer the question:

Is getting a PET scan riskier for ICU patients than a regular CT scan?

All patients in this study will continue to receive their usual critical care. Researchers will closely monitor the scanning process to evaluate its safety.

PET scans are already widely used to detect cancer, but new advancements may allow us to use them more often to diagnose infections. Before this can become routine practice, we need to ensure that PET scanning is just as safe as other commonly used imaging techniques. This study will assess all ICU patients undergoing a PET scan-regardless of the reason for the scan-to determine how safe the procedure is in critically ill individuals.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving PET/CT during ICU admission (any indication)
* Patients undergoing CT Thorax/Abdomen (matched cohort)

Exclusion Criteria:

* CT-scan for any acute indication (acute danger to vital parameters).
* CT-Cerebrum
* Registrion in the dutch Objection to medical research registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients admitted to the Intensive Care Unit (ICU) will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Measured during the transport phase and 4 hours after return to the Intensive Care Unit.
  All adverse events associated with imaging procedures (PET and CT) This will encompass (amongst others) oxygen desaturation, bronchospasm, accidental extubation, hypo-/hypertension, cardiac arrest, malfunctioning medical devices, lack of necessary medication etc.)
  Timeframe: Start transport to PET/CT scanner and 4 hours hands-off time.
  We will score the noted adverse events in a grading scale adapted from the Clavien-Dindo classification that surgeons use to grade the severity of post-operative complications.

SECONDARY OUTCOMES:
Employee dosimetry | Transport and the hands-off time after scan (i.e. 4h in case of [18]FDG PET scanning)
  With regards to radiation protection all medical personnel involved in the (PET) procedure will wear electronic personal dosimetry device to ensure they fall into risk categories as outlined by law.
  Timeframe: Start at injection of radiopharmaceutical for 4 hours (=hands-off period)
Dietary Adjustment | 24-48 hours before scan procedure and until 24 hours after cessation of the diet.
  The effect of the application of dietary adjustments (Ketogenic diet or fasting) on patient safety. Evaluating the incidence of hypertriglyceridemia, pancreatitis and hypo-/hyperglykemia in both patient groups.
  Timeframe: Initiation of preparatory diet for PET-scan. Normally 24 hours - 48 hours before scan until 24 hours after cessation of the diet.
Kidney failure (KDIGO) | Day of the scan and up to 3 days after the scan to evaluate the effect on kidney function (i.e. creatinine and urine creatinine will be measured 4 times and evaluated for significant alterations after the application of iodine contrast (if given))
  To evaluate the incidence of kidney failure when I.V. contrast is applied. Serum creatinine and 24 hours urine creatinine will be checked to estimate clearance

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie the results in the publication will be made available upon request by other researchers.
Supporting Information: Study Protocol
Time Frame: Once data collection has been completed, data will be made available on request. Ergo circa April 2027.
Access Criteria: Only data gathered to answer the primary research question posed in this study will be made available and only upon request via the primary researcher.

REFERENCES:
- [Background] Baldetti L, Busnardo E, Pazzanese V, Ricchetti G, Barone G, Sacchi S, Calvo F, Gramegna M, Pieri M, Ingallina G, Camici PG, Ajello S, Scandroglio AM. Myocardial viability assessment during Impella support with 18-fluorodesoxyglucose PET imaging. ESC Heart Fail. 2025 Feb;12(1):683-687. doi: 10.1002/ehf2.15053. Epub 2024 Sep 6. PMID 39239887
- [Background] Slart RHJA, Tsoumpas C, Glaudemans AWJM, Noordzij W, Willemsen ATM, Borra RJH, Dierckx RAJO, Lammertsma AA. Long axial field of view PET scanners: a road map to implementation and new possibilities. Eur J Nucl Med Mol Imaging. 2021 Dec;48(13):4236-4245. doi: 10.1007/s00259-021-05461-6. Epub 2021 Jun 16. PMID 34136956
- [Background] Schwebel C, Clec'h C, Magne S, Minet C, Garrouste-Orgeas M, Bonadona A, Dumenil AS, Jamali S, Kallel H, Goldgran-Toledano D, Marcotte G, Azoulay E, Darmon M, Ruckly S, Souweine B, Timsit JF; OUTCOMEREA Study Group. Safety of intrahospital transport in ventilated critically ill patients: a multicenter cohort study*. Crit Care Med. 2013 Aug;41(8):1919-28. doi: 10.1097/CCM.0b013e31828a3bbd. PMID 23863225
- [Background] Bercault N, Wolf M, Runge I, Fleury JC, Boulain T. Intrahospital transport of critically ill ventilated patients: a risk factor for ventilator-associated pneumonia--a matched cohort study. Crit Care Med. 2005 Nov;33(11):2471-8. doi: 10.1097/01.ccm.0000185644.54646.65. PMID 16276168
- [Background] Parmentier-Decrucq E, Poissy J, Favory R, Nseir S, Onimus T, Guerry MJ, Durocher A, Mathieu D. Adverse events during intrahospital transport of critically ill patients: incidence and risk factors. Ann Intensive Care. 2013 Apr 12;3(1):10. doi: 10.1186/2110-5820-3-10. PMID 23587445
- [Background] Waydhas C. Intrahospital transport of critically ill patients. Crit Care. 1999;3(5):R83-9. doi: 10.1186/cc362. Epub 1999 Sep 24. PMID 11094486
- [Background] Murata M, Nakagawa N, Kawasaki T, Yasuo S, Yoshida T, Ando K, Okamori S, Okada Y. Adverse events during intrahospital transport of critically ill patients: A systematic review and meta-analysis. Am J Emerg Med. 2022 Feb;52:13-19. doi: 10.1016/j.ajem.2021.11.021. Epub 2021 Nov 20. PMID 34861515
- [Background] Venkategowda PM, Rao SM, Mutkule DP, Taggu AN. Unexpected events occurring during the intra-hospital transport of critically ill ICU patients. Indian J Crit Care Med. 2014 Jun;18(6):354-7. doi: 10.4103/0972-5229.133880. PMID 24987233
- [Background] Brunsveld-Reinders AH, Arbous MS, Kuiper SG, de Jonge E. A comprehensive method to develop a checklist to increase safety of intra-hospital transport of critically ill patients. Crit Care. 2015 May 7;19(1):214. doi: 10.1186/s13054-015-0938-1. PMID 25947327
- [Background] van Leer B, van Rijsewijk ND, Nijsten MWN, Slart RHJA, Pillay J, Glaudemans AWJM. Practice of 18F-FDG-PET/CT in ICU Patients: A Systematic Review. Semin Nucl Med. 2023 Nov;53(6):809-819. doi: 10.1053/j.semnuclmed.2023.05.003. Epub 2023 May 29. PMID 37258380
- [Background] van Snick JH, van Leer B, Nijsten MWN, Pillay J, Slart RHJA, Glaudemans AWJM, van Rijsewijk ND. Long axial field of view PET/CT in critically ill patients: lessons from a case report. Front Med (Lausanne). 2024 Jan 4;10:1347791. doi: 10.3389/fmed.2023.1347791. eCollection 2023. PMID 38239612